CLINICAL TRIAL: NCT01680731
Title: 3-Dimension Ultrasound Findings in Women Who Have Undergone Vacuum Versus Forceps-Assisted Vaginal Deliveries
Brief Title: 3D Ultrasound in Women With Vacuum or Forceps Deliveries
Acronym: VADUS
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Tulin Ozcan MD, Associate Professor of Obstetrics and Gynecology, University of Rochester
Other Study IDs: 39146
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Pelvic Floor Injury; Urinary Incontinence; Stool Incontinence
Keywords: Pelvic floor injury; Levator ani muscle
MeSH Terms: conditions — Urinary Incontinence; Encopresis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Forceps assisted vaginal delivery: Forceps assisted vaginal delivery within 1-5 years without any interval delivery
- Vacuum assisted vaginal delivery: Vacuum assisted vaginal delivery within 1-5 years without any interval delivery
- Elective cesarean delivery: Elective cesarean vaginal delivery within 1-5 years without any interval delivery done prior to labor
- Spontaneous vaginal delivery: Spontaneous vaginal delivery within 1-5 years without any interval delivery

SUMMARY:
The purpose of this study is to investigate of the differences in pelvic floor anatomy and function in women who have undergone a vacuum assisted vaginal delivery (VAVD) versus a forceps assisted vaginal delivery (FAVD) using three-dimensional ultrasound imaging. Women within 1-5 years after first delivery who did not have an internal delivery will be included. The total number of subjects is forty. This will include ten primiparous subjects who have undergone vacuum delivery, ten who have undergone forceps delivery, ten who had spontaneous vaginal delivery and ten who have undergone primary elective cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Females age >18 and <45.
* Primiparous females with singleton pregnancy who have undergone a term vacuum assisted vaginal delivery, forceps assisted vaginal delivery, spontaneous vaginal delivery, or elective primary cesarean section or spontaneous vaginal delivery.
* Birth weight >2500g and <4500g.
* Delivery should have occurred more than one year ago, but less than five years ago.

Pregestational BMI <35kg40kg/m2.

Exclusion Criteria:

* Presence of interim delivery.
* Presence of both vacuum and forceps use during delivery.
* Presence of pregestational or A2 gestational diabetes mellitus.
* Presence of neuromuscular disorder (i.e., spinal cord disease, Multiple Sclerosis, Myasthenia Gravis) or connective tissue disorder (i.e., Lupus and Sjogren's disease).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Forty primiparous subjects with a history of a singleton pregnancy who have undergone a term vacuum assisted vaginal delivery, forceps assisted vaginal delivery, spontaneous vaginal delivery, or elective primary cesarean section or spontaneous vaginal delivery with 10 subjects in each group.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Levator ani injury on 3D ultrasound | 1-5 years after delivery
  Assessment of levator ani injury on trasnperineal 3D ultrasound images

CONTACTS AND LOCATIONS:
Overall Officials: Tulin Ozcan, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States